CLINICAL TRIAL: NCT04427449
Title: Multi-center Phase I/II Clinical Trial of 4SCAR-CD44v6 T Cells for Treating Cancer
Brief Title: 4SCAR-CD44v6 T Cell Therapy Targeting Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Collaborators: Shenzhen Hospital of Southern Medical University (Other); The Seventh Affiliated Hospital of Sun Yat-sen University (Other); Shenzhen Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Lung-Ji Chang, President, Shenzhen Geno-Immune Medical Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-20004
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Cancers Which Are CD44v6 Positive
Keywords: CAR-T; CD44v6; Breast cancer; Gastric cancer; Lymphoma
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms; Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Single arm 4SCAR-CD44v6 T cells to treat cancer (Experimental)
  Interventions: Biological: CD44v6-specific CAR gene-engineered T cells

INTERVENTIONS:
Biological: CD44v6-specific CAR gene-engineered T cells — 4SCAR-CD44v6 Infusion of 4SCAR-CD44v6 T cells at 10^6 cells/kg body weight

SUMMARY:
The purpose of this clinical trial is to assess the feasibility, safety and efficacy of 4SCAR-CD44v6 T-cell therapy targeting multiple cancers. The study also aims to learn more about the function of the CD44v6 CAR-T cells and their persistency in the patients.

DETAILED DESCRIPTION:
CD44 variant domain 6 (CD44v6) which belongs to CD44 family has been implicated in tumorigenesis, tumor cell invasion and metastasis. The expression of CD44v6 was reported for the majority of squamous cell carcinomas, a proportion of adenocarcinomas of differing origin, a proportion of melanoma and lymphoma. This expression pattern has made CD44v6 an attractive target for the therapy of various types of CD44v6 positive cancers.

The T cells from patients or transplantation donors will be genetically modified with lentiviral CAR vector to recognize specific molecules - CD44v6 expressed on the surface of the cancer cells. The engineered T cells will be applied to patients through intravenous delivery.

The purpose of this clinical trial is to assess the feasibility, safety and efficacy of CD44v6 CAR-T cell therapy in multiple cancers including - but not limited to - stomach cancer, breast cancer, prostate cancer, multiple myeloma and lymphoma which are CD44v6 positive. Another goal of the study is to learn more about the function of the 4SCAR-CD44v6 T cells and their persistency in the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age older than 6 months.
2. Confirmed expression of CD44v6 in tumor specimens by immuno-histochemical staining or flow cytometry.
3. Karnofsky performance status (KPS) score is higher than 70 and life expectancy > 3 months.
4. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements: cardiac ejection fraction ≥ 50%, oxygen saturation ≥ 90%, creatinine ≤ 2.5 × upper limit of normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × upper limit of normal, total bilirubin ≤ 2.0mg/dL.
5. Hgb≥80g/L.
6. No cell separation contraindications.
7. Abilities to understand and the willingness to provide written informed consent.

Exclusion Criteria:

1. Sever illness or medical condition, which would not permit the patient to be managed according to the protocol, including active uncontrolled infection.
2. Active bacterial, fungal or viral infection not controlled by adequate treatment.
3. Known HIV, hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
4. Pregnant or nursing women may not participate.
5. Use of glucocorticoid for systemic therapy within one week prior to entering the trial.
6. Receive treatment related to CD44v6 targeted therapy.
7. Patients, in the opinion of investigators, may not be able to comply with the study.

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of infusion | 1 year
  Treatment-related adverse events are assessed by NCI CTCAE V4.0 criteria.
Clinical response | 1 year
  Objective responses (complete response (CR) + partial response (PR)) are assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Shenzhen Children's Hospital, Shenzhen, Guangdong
  - Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong
  - Shenzhen Hospital of Southern Medical University, Shenzhen, Guangdong
  - The Seventh Affilliated Hospital, Sun Yat-Sen University, Shenzhen, Guangdong